CLINICAL TRIAL: NCT00753155
Title: Prospective Intervention Study to Improve HRQoL and Exercise Tolerance After Lnug Transplantation
Brief Title: Prospective Intervention Study to Improve HRQoL and Exercise Tolerance After Lung Transplantation (Ergo-LTx)
Acronym: Ergo-LTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Kugler, Christiane, PhD, Hannover Medical School, Hannover
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LTx-2778
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Lung Transplantation
Keywords: HRQoL;; exercise; capacity
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise training; psychosocial support — supervised home-based endurance training; recommendation to exercise every other day; psychosocial support

SUMMARY:
A prospective, interventional rehabilitation program was initiated to improve exercise capacity and psychosocial functioning in patients after lung transplantation (LTx) and to evaluate long-term effects on health-related quality of life (HRQoL).

Study subjects were randomized to either intervention or to control group and were followed with regular cardiopulmonary exercise testings and HRQoL measurements (SF-36) for 36±3 months after LTx. Patient characteristics did not differ concerning age, gender, and diagnosis at study entry. IG patients received regular psychosocial support and performed a home-based supervised ergometer training program. CG patients were recommended to perform regular exercising.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant (single, double, combined heart-lung) (6-9 mts post Tx)
* Stable health condition at study entry (pt stays within home environment)
* Age ≥ 18 yrs
* Sufficient language skills to answer questionnaire
* Follow-up at our center
* Willingness to participate by written informed consent

Exclusion Criteria:

* BOS III diagnosis before study inclusion
* Episodes of recurrent acute rejections
* Medical contra-indication for regular exercise ergometer training
* Malignancy
* Multi-resistent pathogens

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2002-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
HRQoL, exercise capacity | 36 mts

SECONDARY OUTCOMES:
Weight gain; Pulmonary function; Social re-integration | 36 mts

REFERENCES:
- [Derived] Gutierrez-Arias R, Martinez-Zapata MJ, Gaete-Mahn MC, Osorio D, Bustos L, Melo Tanner J, Hidalgo R, Seron P. Exercise training for adult lung transplant recipients. Cochrane Database Syst Rev. 2021 Jul 20;7(7):CD012307. doi: 10.1002/14651858.CD012307.pub2. PMID 34282853